CLINICAL TRIAL: NCT07348302
Title: Prospective, Randomised, DBPC, Multicenter Clinical Trial to Evaluate Efficacy and Safety of Sublingual Immunotherapy in Patients With Rhinitis/Rhinoconjunctivitis With or Without Mild to Moderate Asthma, Allergic to Dpt and/or Df
Brief Title: Efficacy and Safety of SLIT in Patients With Rhinitis/RC With/Without Mild-moderate Asthma, Due to Dpt and/or Df
Acronym: Oraltek-58
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MM09-SLG-058
Record Dates: First submitted 2025-12-05; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Rhinitis; Rhinoconjunctivitis
Keywords: immunotherapy; sublingual; Quality of live; dust mites; Dermatophagoides pteronyssinus; Dermatophagoides farinae; moderate asthma; allergic rhinitis; Allergic asthma; House dust mite allergy; efficacy; safety
MeSH Terms: conditions — Rhinitis; Rhinitis, Allergic; Dust Mite Allergy | interventions — Desensitization, Immunologic

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, double-blind, placebo-controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Is a solution identical in composition to the active treatment, but without active ingredients
  Interventions: Biological: Allergen Immunotherapy Extract
- Sublingual MM09 (Experimental): Active substance
  Interventions: Biological: Allergen Immunotherapy Extract

INTERVENTIONS:
Biological: Allergen Immunotherapy Extract — Sublingual spray, solution
  Other Names: ORALTEK®

SUMMARY:
The goal of this clinical trial is to learn if MM09 works to treat patients allergic to house mites, displaying rhinitis/rhinoconjunctivitis with or without mild to moderate asthma. It will also learn about the safety of MM09. The main questions it aims to answer are:

Does MM09 reduce the symptoms and the need of rescue medication? What medical problems do participants have when inhaling MM09? Researchers will compare MM09 to a placebo (a look-alike substance that contains no drug) to see if MM09 works to treat rhinitis/rhinoconjunctivitis.

DETAILED DESCRIPTION:
Sublingual MM09 is being investigated as an etiological treatment for moderate-to-severe allergic rhinitis and/or rhinoconjunctivitis (as classified by ARIA), with or without mild-to-moderate controlled allergic asthma (as defined by GINA 2022), caused by Dermatophagoides pteronyssinus and/or Dermatophagoides farinae. This prospective, randomized, double-blind, placebo-controlled, multicenter phase III clinical trial aims to assess the efficacy of sublingual MM09 at a dose of 30,000 TU/mL compared to placebo, administered over 12 months, in participants aged 12 to 65 years.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have signed and dated Informed Consent Form (ICF).
2. Female or male aged 12 to 65 years, both included, at the time of signature of ICF.
3. Participants with confirmed clinical history of inhalation allergy with intermittent or persistent moderate-severe rhinitis/ rhinoconjunctivitis according to the ARIA classification(1) of at least 1 year of duration (treated with anti-allergic medication) with or without mild-moderate controlled intermittent or persistent asthma according to the definition of GINA 2022(2) caused by Dermatophagoides pteronyssinus and/or Dermatophagoides farinae.
4. Participants with positive skin prick test and a wheal major diameter ≥ 5 mm to a standardized allergen extract of Dermatophagoides pteronyssinus and/or Dermatophagoides farinae.
5. Women of childbearing age (i.e., following menarche and until postmenopause, defined as no menses for 12 months without an alternative medical cause, or non-subject to permanent sterilisation methods, such as hysterectomy, bilateral salpingectomy and bilateral oophorectomy) must have a serum pregnancy test negative result, and a confirmed menstrual period before enrolling the study.
6. Women of childbearing age must commit to using a highly effective contraception method during the trial and up to 1 month after the end of treatment with the investigational medicinal product (IMP). Such methods include: combined (estrogen and progestogen containing) hormonal, contraception. associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device, intrauterine hormone-releasing system, male condom, diaphragm used with spermicide, bilateral tubal occlusion, vasectomized partner or sexual abstinence.
7. Participants capable of complying with dosage regimen.
8. Participants owning a smartphone to register symptoms and medication consumption.
9. Participants not sensitized to any other clinically relevant allergen or sensitized with the following characteristics (sensitization to other allergens will be assessed through skin prick test in Europe and LATAM and through IgE levels in China):

   1. Participants sensitized to dander (with a positive skin prick test for dander or IgE ≥ 0.35 kU/L), provided that they have occasional exposure and symptoms.
   2. Participants sensitized to endemic pollen (with a positive skin prick test or IgE ≥0.35 kU/L) will be scheduled to be included so that the pollen season does not coincide with the Baseline Evaluation Period nor with one month before and after the Main Evaluation Period. In LATAM, grass sensitized participants will not be included.
10. Participants not sensitized to moulds, cockroach, Blomia tropicalis or other geographically relevant mites (negative skin prick test or IgE < 0.7 kU/L).
11. Participants with a RCSMS ≥ 3 out of 6 recorded for at least 10 days during the baseline evaluation period, corresponding to moderate-to-severe allergic rhinitis/rhinoconjunctivitis.
12. Participants with specific IgE against a complete extract of D. pteronyssinus and / or D. farinae or any of the molecular components of allergenic sources with a value ≥ 3.5kU/L.

Exclusion Criteria:

1. Participants who have received previous immunotherapy to any of the tested allergen during the last 5 years or any desensitization process in the last 2 years (e.g., oral immunotherapy [OIT], milk, or egg) before the second screening visit (S2), or currently receiving immunotherapy with any other allergen.
2. Those cases in which allergen-specific immunotherapy (AIT) would be a contraindication according to the criteria of European Allergy and Clinical Immunology Immunotherapy Subcommittee.(3)
3. Asthmatic participants with forced expiratory volume in the first second (FEV1) <80% (following at least a 6-hour washout of short-acting beta2 agonists [SABA] and 12-hour washout of long-acting beta2 agonists [LABA]) despite pharmacological treatment by the time of enrolment.
4. Participants with uncontrolled asthma, according to GINA 2022,(2) asthma with poor symptom control (frequent symptoms or reliever use, activity limited by asthma, night waking due to asthma) and/or frequent exacerbations (≥2/year) requiring oral corticosteroids (OCS), or serious exacerbations (≥1/year) requiring hospitalization.
5. Participants with severe asthma, according to GINA 2022,(2) on Step 4 or 5 treatment, who had poor symptom control and had good adherence and inhaler technique.
6. Participants on treatment with β-blockers or angiotensin-converting enzyme (ACE) inhibitor.
7. Participants on treatment with immunosuppressive or biological drugs.
8. Participants who had not had a long enough washout/withdrawal period at the first screening visit (S1) according to criteria in the study protocol (See Table 6 in section 9.5.3) before undergoing allergen diagnostic tests (skin prick test or IgE analysis).
9. Unstable participants who have suffered a respiratory tract infection and/or asthma exacerbation within 4 weeks prior to first screening visit (S1).
10. Participants who have suffered chronic urticaria, severe anaphylaxis, or with hereditary angioedema history within 2 years prior to the first screening visit (S1).
11. Participants having any contraindication for the use of adrenaline (e.g., hyperthyroidism, heart disease, or hypertension) according to the investigator's criteria.
12. Participants with other severe diseases not related to allergic rhinitis or asthma that could interfere with the study treatment or the follow-up.
13. Participants with severe and unresponsive to treatment autoimmune diseases (e.g., thyroiditis or lupus), tumoral diseases or immunodeficiencies.
14. Participants that could not comply with the study protocol, according to the investigator's criteria, or have a serious mental illness.
15. Participants with known allergy to any of the components of the study treatment other than study allergens.
16. Participants who had a complication(s) of any nasal disease (including nasal polyp, nasal septal deviation, and hypertrophic rhinitis, drug-induced rhinitis and/or non-allergic rhinitis) affecting an appropriate evaluation of the efficacy and/or safety, according to investigator's criteria.
17. Participants who had a nasal surgery within 6 months prior to the first screening visit (S1) or have programmed or anticipated nasal surgery during the trial period.
18. Participants with a lesion in the oral cavity that could confound the safety profile of the study treatment, according to the investigator's criteria.
19. Participants who required treatment with antihistamines and/or corticosteroids for other purposes than alleviating symptoms of allergic rhinitis (except temporal use for diseases such as common colds).
20. Participants with lower respiratory tract diseases different from asthma as emphysema, bronchiectasis, or chronic obstructive pulmonary disease.
21. Breastfeeding or pregnant women.
22. Participants who are immediate family members of the investigator.
23. Concurrent participation in other clinical trials or previous participation within 30 days prior to the first screening visit (S1).
24. Participants with history of serious systemic reactions, including food, Hymenoptera venom, medications, etc.
25. Participants expected to have marked changes (e.g., moving) in the circumstances of life during the study.
26. Participants who plan to start using anti-mite bedding or similar equipment during the study.
27. Participants who are considered inappropriate for the study, according to the investigator criteria.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 736 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2029-04-27 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
RCSMS : Rhinitis/Rhinoconjunctivitis Combined Symptom and Medication Score | last 4 weeks of IMP treatment
  The RCMS corresponds to the sum of Rhinitis/Rhinoconjunctivitis Symptom Score (RSS) and Rhinitis/Rhinoconjunctivitis Medication Score (RMS).
  The daily RCSMS will be calculated as RCSMS (0-6) = RSS (0-3) + RMS (0-3)
  Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
RSS : Rhinitis/Rhinoconjunctivitis Symptom Score | last 4 weeks of IMP treatment
  The RSS will correspond to the sum of the grade of the six Rhinitis Rhinoconjunctivitis symptoms score (SS) divided by six:
  RSS (0-3) = (SS1+SS2+SS3+SS4+SS5+SS6) /6. The final RSS will range from 0 to 3.
  Each symptom will be graded 0-3 as follows:
  * 0 = No symptoms (no obvious symptoms).
  * 1 = Mild symptoms (trivial; the symptom is clearly present but not bothersome).
  * 2 = Moderate (annoying but not disabling or intolerable).
  * 3 = Severe (disabling and/or intolerable).
RMS : Rhinitis/Rhinoconjunctivitis Medication Score | last 4 weeks of IMP treatment
  The rhinitis/rhinoconjunctivitis rescue medication will be provided to the participants with the instruction to use them according to a specific stepwise standardised procedure (See section 8.6.2):
  * 0= no medication.
  * 1= if symptoms occur, first take an oral antihistamine (desloratadine) with or without ocular antihistamine (olopatadine)
  * 2= if symptoms are insufficiently controlled, add intranasal corticosteroid (INS) with or without oral antihistamine (fluticasone furoate).
  * 3= if symptoms persist and are insufficiently controlled add an oral corticosteroid (OCS) (methylprednisolone) (with or without intranasal corticosteroid [INS] and antihistamine)
ASS : Asthma Symptom Score | last 4 weeks of IMP treatment
  The score is obtained by the collection on the occurrence of following asthma symptoms:
  * Cough
  * Wheezing
  * Shortness of breath or feeling of choking
  * Chest tightness
  Each asthma symptom will be graded as follows:
  * 0= No symptoms (no obvious symptoms).
  * 1= Mild symptoms (trivial; the symptom is clearly present but not bothersome).
  * 2= Moderate (annoying but not disabling or intolerable).
  * 3= Severe (disabling and/or intolerable).
  The ASS will correspond to the sum of the grades of the four asthma symptoms score (SS) divided by four:
  ASS (0-3) = (SS1+SS2+SS3+SS4) /4. The final score will range from 0 to 3.
AMS: Asthma Medication Score | last 4 weeks of IMP treatment
  The AMS will be scored based on the therapeutic step in which the drugs are included in the GEMA 5.0 (90) and GINA 2020 guidelines.(91) The scoring method is detailed in the article entitled "Combination of Allergic Asthma Symptom and Medication Scores in Allergen Immunotherapy Trials: A Proposal."
  The steps of medication shown in the Figure 6 (above) correspond to the medication stepping of GEMA 5.0. In asthma participants AMS will be score as follows:
  * 0.5= SABA as needed.
  * 1= Low dose ICS with/without SABA as needed.
  * 1.5= Low dose ICS + LABA or medium dose ICS with/without SABA as needed.
  * 2= Medium dose ICS+LABA with/without SABA as needed.
  * 2.5= High dose ICS+LABA with/without SABA as needed.
  * 3= High dose ICS+LABA + systemic corticosteroids with/without SABA as needed. The AMS will correspond to the highest level of medication taken on a day. The score will range from 0 to 3.
ARSS: Asthma and Rhinitis/Rhinoconjunctivitis Symptom Score | last 4 week of IMP treatment
  The ARSS ranges from 0 to 6, corresponds to the sum of RSS and ASS, and is calculated as follows: ARSS (0-6) = RSS (0-3) + ASS (0-3)
  Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Caballero, Study Chair — Inmunotek S.L.
Locations (19):
- Argentina (6):
  - Centro Médico Vitae, Nueve de Julio, Buenos Aires
  - Centro de Investigaciones Clínicas - Instituto de Especialidades de la Salud Rosario, Rosario, Santa Fe Province
  - Centro Respiratorio Infantil, Rosario, Santa Fe Province
  - Fundación CIDEA, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Centro de Educación Medica de Investigaciones Clinicas "Norberto Quirno" (CEMIC), Buenos Aires
- China (9):
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - The Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Zhongshan, Guangzhou
  - The Third Xiangya Hospital of Central South University, Xiangya, Hunan
  - Changzhou Third People's Hospital, Changzhou, Jiangsu
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Tongji Hospital Tongji Medical College of HUST, Tongji, Wuhan
  - Union Hospital Tongji Medical College of HUST, Huangzhou
- Portugal (2):
  - Unidade de Local de Saúde de Santo António, E.P.E., Porto
  - ULS Lezíria- Hospital Distrital de Santarém, Santarém
- Spain (2):
  - Hospital IMED Benidorm, Benidorm, Alicante
  - Hospital General Universitario Dr. Balmis, Alicante

IPD SHARING:
Plan to Share IPD: No